CLINICAL TRIAL: NCT06455241
Title: Feasibility and Efficacy of HABIT - a Novel Occupational Therapy Intervention for Enhancing Daily-Use of the Affected Upper Extremity Among Individuals Post Stroke.
Brief Title: Feasibility and Efficacy of HABIT for Enhancing Daily Hand-Use Post Stroke
Acronym: HABIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Debbie Rand, Associate Professor, Researcher at department of occupational therapy, Head of 'Gaming for Rehabilitation' Lab, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HABIT 0008389-4
Record Dates: First submitted 2024-06-01; First posted 2024-06-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Self-efficacy; Behavior; Stroke; Group intervention; Daily Hand-use
MeSH Terms: conditions — Stroke; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HABIT (Experimental): All participants will receive HABIT - a novel occupational therapy intervention.
  HABIT will include 10 sessions (2 sessions per week for 5 weeks). HABIT will include small group of 5-8 participants, so approximately 4 rounds of HABIT will be needed to reach 20 participants
  Interventions: Other: HABIT (Hand Activities Behavior Intervention)

INTERVENTIONS:
Other: HABIT (Hand Activities Behavior Intervention) — A Novel Occupational Therapy Intervention for Enhancing Daily Hand-Use of the affected upper extremity Among Individuals post Stroke.

SUMMARY:
This experimental design will assess the feasibility & initial effectiveness of HABIT - a novel occupational therapy to increase the daily hand-use of the affected upper extremity post stroke.

Assessments will be conducted at four time points: baseline, pre, post the HABIT intervention and follow-up (by phone) .

DETAILED DESCRIPTION:
The goal of this study is to test the feasibility and efficacy of HABIT (Hand Activities Behavior Intervention) in increasing daily hand-use of the affected upper extremity among individuals with good motor ability post-stroke.

The aim of HABIT is to increase the daily use of the weaker hand in everyday activities by improving non-motor components (such as self-efficacy, raising the frustration threshold for performing tasks with the affected upper extremity, and creating opportunities for hand use). HABIT will include group discussions, analysis of challenges in using the affected upper extremity, home exercises, problem-solving and practice and dual-task activities. The intervention will focus on raising awareness, changing habits, and practicing the use of the affected upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above residing in their own homes
* Hebrew speakers
* Up to 10 years post-stroke
* Mild upper extremity motor impairment but still report difficulty using their hand. This will be determined by a total score of 43/66, including the Hand subtest score of 7/14 points of the Fugl-Meyer Motor Assessment.
* No significant cognitive decline (score of 19 and above on Montreal Cognitive Assessment)
* Able to walk with or without assistive devices
* Able to provide informed consent by signing a consent form
* Full function of both hands and independent in daily function prior to stroke

Exclusion Criteria:

* Other neurological conditions or psychiatrists
* with moderate or significant proprioception deficit (Thumb Localization Test >1)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in scores of the Rating of Everyday Arm-Use in the Community and Home (REACH) | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week) and change from post to follow-up (3-6 months)
  A short questionnaire assessing the level of daily use of the affected hand after stroke in daily activities. The questionnaire consists of 2-5 questions (depending on the responses being assessed), from which a score is obtained determining the level of use of the affected hand. The score ranges from 0 (no use of the affected hand) to 5 (full use).
Change in scores of the Canadian Occupational Performance Measure (COPM) | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week) and change from post to follow-up (3-6 months)
  Change in scores of performance and satisfaction of performance for therapeutic goals that the participants define as important to them. Goals will focus on using the affected upper extremity.

SECONDARY OUTCOMES:
Change in Upper-Extremity-Cognitive Dual Task capacity | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week)
  The dual-task will include the Box and Block test (number of blocks transferred in one minute) and the counting backward task in increments of 3 from a three-digit number (number of correct answers in one minute).
Change in Confidence in Arm and Hand Movement scale (CAHM) | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week) and change from post to follow-up (3-6 months)
  This is a 20-item questionnaire assess the self-efficacy to use the affected hand after stroke in social, household, and community contexts.
Satisfaction from the HABIT intervention | post intervention (week 8) and at follow-up (3-6 months by phone)
  A self-report questionnaire assessing the satisfaction with the novel intervention
Change in Upper-extremity Motor Activity Log (UE-MAL) | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week) and change from post to follow-up (3-6 months)
  This instrument is a structured interview intended to examine how much and how well the subject uses their more-affected arm outside of the laboratory setting. Participants are asked standardized questions about the amount of use of their more-affected arm (Amount Scale or AS) and the quality of their movement (How Well Scale or HW) during the functional activities indicated. The scales are printed on separate sheets of paper and are placed in front of the participant during test administration. participants should be told that they can give half scores (i.e., 0.5,1.5,2.5,3.5,4.5) if this is reflective of their ratings. 0-not used to 5- same as pre-stroke/ normal.
Change in U-rate UE | no change from baseline (0 week) to pre intervention (3 week) but change from pre to post intervention (8 week) and change from post to follow-up (3-6 months)
  U-Rate-UE includes the following single self-perceived question: "please rate how much your affected UE has recovered from your stroke ". Participants were presented with a 10- point vertical scale starting at the bottom from 0 (no recovery) to 100 (full recovery) at the top of the scale but could rate any whole number from 0 to 100. Participants were asked to rate this question verbally or by pointing on the scale to estimate the extent to which the affected UE has recovered from the stroke as a percentage of its full(pre stroke) ability.

OTHER OUTCOMES:
Demographic and stroke information questionnaire | baseline (week 0)
  to describe the participants
Functional Independence Measure | baseline (week 0)
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations. It includes 18-items of basic activities. Each item in rated from 1 (not independent) to 7 (independent) points. The total score for the FIM instrument will be a value between 18 and 126.
Instrumental Activities of Living (IADL) questionnaire | baseline (week 0) and at follow-up (3-6 months)
  to assess independence in IADL
Thumb localization test TLT | baseline (week 0)
  This is a standard assessment for evaluating proprioceptive sensation in individuals after a stroke. With the participant's eyes closed, the examiner moves the affected hand into four different positions. The participant is then required to grasp the thumb of the affected hand with their strong hand. The ability to grasp the thumb in each of the positions is rated from 0 (normal) to 3 (significant sensory impairment). The final score of the assessment is the lowest score among the four positions.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Rand, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachar Kirshenboim Y, Levy A, Rand D. The hand activity and behavior intervention (HABIT): a novel group to increase daily hand-use post-stroke. Disabil Rehabil. 2026 Jan 4:1-14. doi: 10.1080/09638288.2025.2609762. Online ahead of print. PMID 41485200